CLINICAL TRIAL: NCT02994719
Title: Gait Pattern Analysis in Neurological Disease
Brief Title: Gait Analysis in Neurological Disease
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Veronique Vanderhorst, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2015P000310
Record Dates: First submitted 2015-12-21; First posted 2016-12-16 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Parkinson's Disease; Parkinsonian Disorders; Atypical Parkinson Disease; Progressive Supranuclear Palsy; Multiple System Atrophy; Corticobasal Degeneration; Gait, Frontal; Huntington Disease
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Parkinson Disease, Familial, Type 1; Supranuclear Palsy, Progressive; Multiple System Atrophy; Corticobasal Degeneration; Gait Disorders, Neurologic; Huntington Disease | interventions — carbidopa, levodopa drug combination; Pramipexole; ropinirole; Amantadine; Tolcapone; entacapone; Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Neurological Disease subjects: Parkinson's Disease and other Parkinsonian Disorders subjects. Other Parkinsonian Disorders include Atypical Parkinsonism such as Progressive Supranuclear Palsy, Multiple System Atrophy, Corticobasal Degeneration, Primary Gait Freezing Disorder, Indeterminate Parkinsonian Syndrome. During the first visit no intervention will take place. There is an optional second visit during which subjects with Parkinson's Disease are asked to come come off antiparkinson medication and if applicable, off both medication and deep brain stimulation.
  Interventions: Drug: Anti-Parkinson medication; Device: Deep Brain Stimulation
- Healthy control subjects: The healthy control subjects will be age- and sex-matched to the Neurological Disease subjects.
- Ataxia Subjects: The ataxia subjects will participate in an additional cohort that will test and validate the gait model.
- Huntington Disease Subjects: The Huntington Disease subjects will participate in an additional cohort that will test and validate the gait model.

INTERVENTIONS:
Drug: Anti-Parkinson medication — During the optional second visit subjects with neurological disease and already on anti-parkinson medication are asked to come off their anti-parkinson medication.
  Other Names: Carbidopa/levodopa; pramipexole; ropinirole; amantadine; tolcapone; entacapone
  Groups: Neurological Disease subjects
Device: Deep Brain Stimulation — During the optional second visit subjects with neurological disease already treated with deep brain stimulation are asked to come temporarily stop deep brain stimulation and resume stimulation, with walking trials done in each condition.
  Groups: Neurological Disease subjects

SUMMARY:
The purpose of this study is to investigate whether speed-dependent measures of gait can be identified in patients with neurological conditions that affect gait, particularly in subjects with parkinsonian disorders.

DETAILED DESCRIPTION:
This study aims to determine whether the gait patterns in these subjects differ in predictable and quantifiable ways from those of age- and sex-matched healthy controls. This will be conducted by asking 40 Parkinsonian disorder subjects and 40 age-matched healthy control subjects to walk 9 trials over an 18 ft walkway embedded with pressure sensors at baseline, self-selected slower and faster speeds. In addition, the protocol aims to investigate whether clusters of gait patterns can be identified within subgroups of individuals with parkinsonian disorders with varying co-morbidities or treatment conditions as well as patients with ataxia syndromes. For this aim an additional 20 Parkinsonian disorder subjects need to be recruited. Patients with parkinsonism as defined by UK PD Brain Bank Criteria (n=60), subjects with acquired or inherited ataxic syndromes (n=10) and age- and sex matched controls (n=40) will be recruited. There is an optional second visit in the protocol during which approximately 20 subjects with Parkinsonian disorders, who are willing to come off antiparkinson medication and if applicable, off both medication and deep brain stimulation, are asked to walk an additional 9 trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 (for both healthy and affected subjects).
* Presence of at least 2 of the following: bradykinesia, rest tremor, rigidity, postural instability (UK PD Brain Bank Criteria) (Affected subjects only).
* Montreal Cognitive Assessment will be employed to determine whether subjects will need the assent of a legally authorized representative. Subjects with MOCA ≤ 21 will be consented only with the assent of the subject and informed consent of the authorized legal representative (Affected subjects only).
* These may include subjects who may have indeterminate parkinsonism, when it is not clear whether they have idiopathic Parkinson's Disease versus one of the Atypical Parkinsonisms, such as Vascular Parkinsonism, Multiple System Atrophy, Progressive Supranuclear Palsy, Normal Pressure Hydrocephalus or Corticobasal Degeneration (Affected subjects only).
* Subjects with assistive devices will be eligible for the study and may use them during the study (Affected subjects only).
* Absence of complaints regarding difficulty walking such as arthritic pain, fatigue during walking or slowness of walking (Healthy subjects only).

Exclusion Criteria:

* Presence of alternative explanation for parkinsonism such as head trauma, drug-induced parkinsonism (affected subjects only).
* Currently being treated for major medical illness requiring recent hospitalization (<14 days) (for both healthy and affected subjects).
* Currently participating in another clinical study with an intervention arm (for both healthy and affected subjects).
* Inability to consent due to cognitive impairment and absence of legally authorized representative (for both healthy and affected subjects).
* Subjects with any cardiac, pulmonary conditions (congestive heart failure requiring hospitalization within the past 90 days, recent myocardial infarction < 90 days, supplemental oxygen-requiring subjects due to cardiac or pulmonary conditions) that limit their ability to safely participate in a walking trial (for both healthy and affected subjects).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with Parkinsonism as defined by UK PD Brain Bank Criteria. The study population includes subjects with Parkinson's Disease and may also include subjects who may have indeterminate parkinsonism, when it is not clear whether they have idiopathic Parkinson's Disease versus one of the Atypical Parkinsonisms, such as Vascular Parkinsonism, Multiple System Atrophy, Progressive Supranuclear Palsy, Normal Pressure Hydrocephalus or Corticobasal Degeneration.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Gait speed | through study completion, an average of 1 year
  Method of assessment: physiological parameter

SECONDARY OUTCOMES:
Swing duration | through study completion, an average of 1 year
  Method of assessment: physiological parameter
Stance duration | through study completion, an average of 1 year
  Method of assessment: physiological parameter
Cadence | through study completion, an average of 1 year
  Method of assessment: physiological parameter
Stride length | through study completion, an average of 1 year
  Method of assessment: physiological parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center BIDMC, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No